CLINICAL TRIAL: NCT01403207
Title: An Analysis of Potential Sex Differences in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Mary O'Connor (Other)
Collaborators: Society of Women's Health Research (Unknown); University of Calgary (Other); Florida State University (Other); Georgia Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Mary O'Connor, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 11-001468
Record Dates: First submitted 2011-07-07; First posted 2011-07-27 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Degenerative Joint Disease; Osteoarthritis
Keywords: Sex differences; knee joint; inflammatory mediators; Vitamin D; osteoarthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- knee osteoarthritis: Many musculoskeletal conditions are impacted by the chromosomal sex of the patient. While osteoarthritis (OA) is predominant in men younger than 50 years of age, after age 50 the condition is more prevalent in women, particularly post-menopause. This has implications for diagnosis and treatment of OA, as well as for joint replacement.
  Interventions: Other: musculoskeletal

INTERVENTIONS:
Other: musculoskeletal — Many musculoskeletal conditions are impacted by the chromosomal sex of the patient. While osteoarthritis (OA) is predominant in men younger than 50 years of age, after age 50 the condition is more prevalent in women, particularly post-menopause. This has implications for diagnosis and treatment of OA, as well as for joint replacement.

SUMMARY:
This pilot study will use tissues and fluids that are normally discarded during the course of total knee replacement surgery to investigate potential sex differences in knee osteoarthritis. Basic clinical demographic information will be obtained as well as preoperative functional and pain assessment scores, functional tests, and pressure pain threshold measurement. The purpose of the study will be to investigate if any sex differences can be identified in these tissues and to investigate if there appears to be any relationship between these differences and functional scores and tests.

DETAILED DESCRIPTION:
The goal of this study is to determine if sex differences can be identified in the knee joint that can contribute to the differences in incidence and severity of knee osteoarthritis observed in men and women, particularly over the age of 50. Recent studies assessing the responses of articular chondrocytes to systemic factors suggest that there are underlying differences in the biochemical and molecular characteristics of male and female cells. It is also known that immune responses differ in males and females, suggesting that there may be important differences in the levels of immune modulators in the joint tissues, including the synovial membrane, the synovial fluid, and the cartilage itself. Responses to the vitamin D metabolite 1_,25(OH)2D3 are upregulated in osteoarthritic cartilage, raising the possibility that males and females differ in their circulating levels of vitamin D, in the content of vitamin D metabolites in the synovial tissues, or in the ability of the cells to respond to this steroid. Similarly, in post-menopausal women, circulating estrogen is reduced relative to testosterone, but it is not known if this might impact the knee. Most importantly, it is not known if potential sex differences can be correlated with severity of disease.

This study is based on the hypothesis that sex differences exist in different tissues of the knee joint, which contribute to the increased incidence and severity of knee osteoarthritis in older women as compared to older men.

To test this hypothesis, the investigators will use tissues and fluids that are normally discarded during the course of total knee replacement surgery to investigate potential sex differences.

ELIGIBILITY:
Inclusion Criteria:

1. Patient demographics (age, sex, BMI). 2. Clinical background material

1. Post menopausal female
2. List of all medications and supplements

   1. Use of vitamin D supplements (duration and amount)
   2. Use of bisphosphonates (past and current)
   3. Use of estrogen (past and current)
3. Prior trauma or knee surgery

   1. Have you ever injured the operative knee so badly that it was difficult for you to walk for at least one week?
   2. Have you ever had any kind of knee surgery? Please include arthroscopy (where they put a scope in your knee), ligament repair surgery, or a meniscectomy (where they repaired or cut away a torn meniscus or cartilage)?
4. Prior intraarticular injections

   1. Steroid
   2. Hyaluronic acid
5. SF 12
6. WOMAC
7. PASE functional scale
8. Pain scale: The 11 question OARSI-OMERACT pain scale will be used. Patients will complete the pain scale within 2 weeks prior to surgery and at 3 months following surgery
9. Knee pain map: Patients will complete this within 2 weeks prior to surgery and at 3 months following surgery
10. Pressure pain thresholds at knee. This will be completed within 2 weeks prior to the surgery and at 3 months following surgery (see attachment for details) 3. Preoperative blood tests

a. Vitamin D level 25 D3 should be measured 4. Standard preoperative radiographs: AP, lateral, standing flexion AP and patellar sunrise

Exclusion Criteria:

1. Patients with inflammatory arthritis
2. Patients with osteonecrosis
3. Patients with prior upper tibial osteotomy
4. Premenopausal women
5. Patients under age 65 years, older than 75 years
6. Patients who are insulin dependent or diabetic
7. Patients with a BMI>30
8. Patients with a history of knee infection

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patient enrollment will consist of 10 females and 10 male patients stratified by age. Enrollment is anticipated to be completed over a 12 month time period. Only non Hispanic White patients will be included in the study. Patients must be between 65 and 75 years of age. Patients with a BMI greater than 30 will be excluded
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine if there are sex-differences in different tissues of the knee joint | 1 year
  1. To determine if there are sex-differences in the presence of inflammatory mediators .
  2. To determine if there are sex-differences in the amounts of vitamin D metabolites,estradiol
  3. To determine if there are sex-differences in the responses of osteoblasts from the subchondral bone and chondrocytes from the OA lesion metabolites, estradiol or testosterone.
  4. To determine if there are sex-differences in the content and distribution of neural markers in synovial tissue, menisci and cartilage.

SECONDARY OUTCOMES:
Analyze preoperative functional and clinical data to determine if there are differences in Vitamin D levels and gender differences. | 1 year
  Analyze preoperative functional and clinical data to determine if there are differences in Vitamin D levels and gender differences.

CONTACTS AND LOCATIONS:
Overall Officials: Mary I O'Connor, MD, Principal Investigator — Mayo Clinic Jacksonville, Chair, Orthopedics
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States